CLINICAL TRIAL: NCT02679274
Title: Cycled Testosterone Therapy to Improve Physical Function in Frail Nursing Home Residents
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Lack of funding.
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 15-0176
Record Dates: First submitted 2015-12-15; First posted 2016-02-10 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-01

CONDITIONS: Aging
Keywords: Aging, Frailty, Hypogonadism
MeSH Terms: conditions — Frailty; Hypogonadism | interventions — Sodium Chloride; Testosterone; testosterone enanthate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo injection (saline) to be received on weeks 0, 1, 4, 5, 8 and 9.
  Interventions: Drug: Placebo
- Testosterone (Experimental): Testosterone Enanthate injections (25mg/injection females; 100mg/injection males) to be received on weeks 0, 1, 4, 5, 8 and 9.
  Interventions: Drug: Testosterone

INTERVENTIONS:
Drug: Placebo — Intermittent intramuscular injections of saline (males and females).
  Other Names: Saline
  Arms: Placebo
Drug: Testosterone — Intermittent intramuscular injections of 100 mg Testosterone Enanthate (males) or 25 mg Testosterone Enanthate (females).
  Other Names: Testosterone Enanthate
  Arms: Testosterone

SUMMARY:
Frailty is a recognized cause for disability, hospitalization, and mortality in nursing home residents. Testosterone treatment is among the potentially beneficial treatments in addition to resistance exercise for improving muscle strength and mass in frail adults. The investigators have demonstrated that cycled administration of testosterone improves muscle mass and strength in healthy adults. It is proposed that cycled testosterone administration may be an effective adjuvant therapy for frail older men and women during rehabilitation programs. The hypothesis is that testosterone treatment in addition to standard-of-care (SOC) rehabilitation will result in improved muscle mass and physical function when compared to patients receiving SOC only. Therefore, in a randomized, double-blind, placebo controlled study, the investigators will test the effects of cycled testosterone administration (2 week on treatment, 2 weeks off treatment) on body composition and physical function in male and female nursing home residents undergoing rehabilitative care. Primary outcomes will be assessed before and after 10 weeks of treatment using bioelectric impedance, handgrip dynamometers, short physical performance battery (SPPB), and quality of life (QOL) questionnaires. Data from this pilot project will become the foundation for the development of a larger long-term project solicitation to the NIH aimed at elucidating the efficacy of testosterone treatment on physical function and independence in frail older adults.

DETAILED DESCRIPTION:
Frailty with aging is a serious debilitating condition that can further contribute to a downward spiraling of health and physical function. Many long term nursing home patients enter into rehabilitative care programs with the intent to increase strength and physical independence. However, many patients have lasting functional limitations despite rehabilitation programs intended to improve their physical function and sarcopenia and frailty is common among nursing home residents. Aging in general, and frailty in particular, has been associated with decreases in sex hormones, and testosterone treatment has known anabolic effects to muscle of hypogonadal as well has eugonadal males. Effective adjuvant treatments that can be safely employed in conjunction with existing therapies such as rehabilitative care intended to improve function can have profound benefits to the long-term outcome of male and female patients.

The investigators have demonstrated that administration of testosterone (100 mg/wk) starts showing improvements in lean body mass (LBM) as early as 4 weeks and muscle strength by 8 weeks in healthy older community dwelling males (Sheffield-Moore et al., 2011). In this study, both continuous weekly treatment as well as intermittent treatment (4 weeks on testosterone, 4 weeks off testosterone, etc) resulted in similar benefits after 20 weeks. In addition, the investigators recently completed a 10-week study where the investigators showed both the safety and efficacy of cycled testosterone treatment (100 mg/wk for 2 weeks, alternated by 2 weeks of no treatment) in combination with regular exercise in healthy eugonadal adult men confined to continuous bed rest (see preliminary data). In that study, testosterone robustly increased LBM in as little as 2 weeks of bed rest and improvements in LBM were associated with better protection of physical function upon reambulation.

It is proposed that a cycled testosterone paradigm may be a safe and effective adjuvant therapy for frail older nursing home patients undergoing physical rehabilitation. The investigators hypothesize that testosterone treatment in addition to standard-of-care (SOC) physical therapy or rehabilitation will result in improved muscle mass and physical function when compared to patients receiving SOC only. The long term goal is to develop effective treatments against the functional declines in muscle mass and strength that contribute to the development and progression of frailty. Therefore, the investigators will test the specific aims outlined below in older male and female residents engaging in rehabilitation care at health care centers in Texas City and Galveston. Men and women (age 60-up) will be recruited as they enroll into rehabilitative care programs, screened upon informed consent, and if eligible, block-randomized (double-blinded) to receive either testosterone enanthate (100 mg/wk for males and 25 mg/wk for females) or placebo (saline) treatment for 10 weeks. The treatment will follow a 2-week cycle (2 weeks on-treatment, 2 weeks off, etc). Primary outcomes will be assessed using non-invasive methods at baseline and at completion of the study after 10 weeks. These outcomes will include body composition as determined with bioelectric impedance analysis (BIA), muscle strength and fatigue by handgrip dynamometry, physical function by a short physical performance battery (SPPB), and quality of life (QOL) by a short battery of questionnaires. Blood samples will be collected at screening for safety and will be repeated at completion of the study for secondary outcome measures (hormones, lipid profiles and blood chemistries).

Specific Aim 1. Determine the effects of cycled testosterone treatment on body composition in male and female nursing home residents undergoing rehabilitative care.

Specific Aim 2. Determine the effects of cycled testosterone treatment on physical function in male and female nursing home residents undergoing rehabilitative care.

Data from this pilot/feasibility project will become the foundation for the development of a larger long-term project solicitation to the NIH aimed at elucidating the efficacy of testosterone treatment on physical function and independence in frail older adults.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female
2. Ages: 60 years or older
3. Starting rehabilitative care

Exclusion Criteria:

1. Inability to perform the functional tests specific to the study protocol
2. Diagnosed with carcinomas of the breast or with known or suspected carcinomas of the prostate.
3. Uncontrolled endocrine or metabolic disease (e.g. liver disease, renal disease, diabetes).
4. Uncontrolled hypertension. Systolic blood pressure =/> 160mm Hg or a diastolic blood pressure =/> 100mm Hg on three consecutive measurements taken at one-week intervals. Testosterone, other anabolic steroids and glucocorticoids can cause fluid retention that could worsen uncontrolled hypertension. Subjects will be included if they are on two or less blood pressure medications and have a blood pressure below these criteria.
5. History of significant liver disorders or a 3-fold elevation of liver function tests (Alk phos, ALT, AST). Testosterone can have hepatotoxic effects in some subjects and should be used with careful monitoring of LFTs (liver function), though injections of testosterone at a 100 mg dose is not typically sufficient to negatively affect LFTs.
6. History of angina that occurs with exertion or at rest or a myocardial infarction within the last 12 months.
7. LDL cholesterol greater than 200 mg/dL as testosterone administration may elevate LDL cholesterol levels further, though this is not anticipated with testosterone injections of 100 mg/wk.
8. Hematocrit greater than 51%.
9. Established chronic obstructive pulmonary disease, or untreated sleep apnea.
10. Implanted artificial pacemaker/defibrillator. BIA uses small currents and is not recommended for participants with a pacemaker.
11. Diagnosed systemic fungal infections.
12. Positive screening for HIV or active hepatitis*.
13. Use of or history of recent anabolic steroid use (within 3 months).
14. Alcohol or drug abuse.
15. Any other condition or event considered exclusionary by the PI and covering faculty physician.
16. Vulnerable populations including: individuals unable to consent on their own behalf, prisoners and pregnant women.

    * Subjects excluded due to positive screening results, including HIV, HBV or HCV, will be immediately scheduled for counseling and follow-up testing as needed, and will be advised to consult their primary physician.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-02-16 (Actual); Primary Completion 2016-09-20 (Actual); Study Completion 2016-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edgar L Dillon, PhD, Principal Investigator — University of Texas Medical Branch (UTMB)
Locations (2):
- United States (2):
  - Gulf Health Care Center, Galveston, Texas
  - Gulf Health Care Center, Texas City, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Testosterone
Started (One (1) subject withdrew after consent, and randomization but before study testing started.) | 2 | 1
Completed | 1 | 1
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Testosterone | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Continuous [Mean (Full Range); unit: years] | 83 [83 to 83] | 65 [65 to 65] | 74 [65 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2
Weight [Mean (Full Range); unit: kg] | 65 [65 to 65] | 96 [96 to 96] | 80 [65 to 96]
Fat Mass [Mean (Full Range); unit: Percent Body Mass] | 31 [31 to 31] | 51 [51 to 51] | 41 [31 to 51]
BMI [Mean (Full Range); unit: kg/m^2] | 27 [27 to 27] | 43 [43 to 43] | 35 [27 to 43]

OUTCOME MEASURES:

1. Primary Outcome: Change in Fat-free Mass as Measured by Bioelectric Impediance Analysis (BIA)
Description: Fat-free Mass (kg) calculated from total weight (kg) and percent body fat (%) obtained during bioelectric impedance analysis (BIA).
Time Frame: 0 to 10 Weeks
Measure: Number; unit: kg
Arm/Group | Placebo | Testosterone
Number analyzed (Participants) | 1 | 1
kg | 0.8 | 2.5

2. Secondary Outcome: Change in Handgrip Strength
Description: Measured using a handgrip dynamometer
Time Frame: 0 to 10 Weeks
Measure: Number; unit: kg
Arm/Group | Placebo | Testosterone
Number analyzed (Participants) | 1 | 1
kg | -5.0 | 5.0

3. Secondary Outcome: Change in Knee Extension Strength (Seated)
Description: Collected using a manual muscle tester (MMT).
Time Frame: 0 to 10 Weeks
Measure: Number; unit: kg
Arm/Group | Placebo | Testosterone
Number analyzed (Participants) | 1 | 1
kg | 1.7 | 5.9

4. Secondary Outcome: Change in Hip Abduction Strength (Supine)
Description: Collected using a manual muscle tester (MMT).
Time Frame: 0 to 10 Weeks
Measure: Number; unit: kg
Arm/Group | Placebo | Testosterone
Number analyzed (Participants) | 1 | 1
kg | 0.9 | 2.6

5. Secondary Outcome: Side by Side Balance as Measured by Short Physical Performance Battery (SPPB) at Baseline
Description: During the Short Physical Performance Battery (SPPB) side by side balance test subjects are asked to stand with their feet together and balance for a maximum of 10 seconds. If they are unable to perform balance test, they receive a score of 0 seconds, maximum score is 10 seconds. A higher score indicates a better outcome.
Time Frame: baseline
Measure: Number; unit: seconds
Arm/Group | Placebo | Testosterone
Number analyzed (Participants) | 1 | 1
seconds | 0 | 10

6. Secondary Outcome: Side by Side Balance as Measured by Short Physical Performance Battery (SPPB) at 10 Weeks
Description: as for outcome 5
Time Frame: 10 Weeks
Measure: Number; unit: seconds
Arm/Group | Placebo | Testosterone
Number analyzed (Participants) | 1 | 1
seconds | 10 | 10

7. Secondary Outcome: Semi-Tandem Balance as Measured by Short Physical Performance Battery (SPPB) at Baseline
Description: During the Semi-Tandem Balance section of the Short Physical Performance Battery (SPPB) subjects are asked to stand with their feet in a semi-tandem stance (heel of one foot placed to side of the first toe of the other foot) and balance for a maximum of 10 seconds. If they are unable to perform balance test, they receive a score of 0 seconds, maximum score is 10 seconds. A higher score indicates a better outcome.
Time Frame: baseline
Measure: Number; unit: seconds
Arm/Group | Placebo | Testosterone
Number analyzed (Participants) | 1 | 1
seconds | 0 | 0

8. Secondary Outcome: Semi-Tandem Balance as Measured by Short Physical Performance Battery (SPPB) at 10 Weeks.
Description: as for outcome 7
Time Frame: 10 Weeks
Measure: Number; unit: seconds
Arm/Group | Placebo | Testosterone
Number analyzed (Participants) | 1 | 1
seconds | 10 | 10

9. Secondary Outcome: Tandem Balance as Measured by Short Physical Performance Battery (SPPB) at Baseline
Description: During the Tandem Balance section of the Short Physical Performance Battery (SPPB) subjects are asked to stand with their feet in a tandem stance (heel of one foot directly in front of the toes of the other foot) and balance for a maximum of 10 seconds. If they are unable to perform balance test, they receive a score of 0 seconds, maximum score is 10 seconds. A higher score indicates a better outcome.
Time Frame: baseline
Measure: Number; unit: seconds
Arm/Group | Placebo | Testosterone
Number analyzed (Participants) | 1 | 1
seconds | 0 | 0

10. Secondary Outcome: Tandem Balance as Measured by Short Physical Performance Battery (SPPB) at 10 Weeks
Description: as for outcome 9
Time Frame: 10 Weeks
Measure: Number; unit: seconds
Arm/Group | Placebo | Testosterone
Number analyzed (Participants) | 1 | 1
seconds | 0 | 2.6

11. Secondary Outcome: Change in Gait Speed as Measured by Short Physical Performance Battery (SPPB).
Description: During the gait speed section of the Short Physical Performance Battery (SPPB) subjects are timed while walking a predefined 4 meter course. Data is shown as change in speed (meters/second) from baseline (0 weeks) to 10 weeks. A increase in speed indicates a better outcome.
Time Frame: 0 to 10 Weeks
Measure: Number; unit: meters/second
Arm/Group | Placebo | Testosterone
Number analyzed (Participants) | 1 | 1
meters/second | 0.10 | 0.48

12. Secondary Outcome: Chair Raise as Measured by Short Physical Performance Battery (SPPB) at Baseline
Description: During the chair rise section of the Short Physical Performance Battery (SPPB), subjects are timed while they rise from a seated (chair) to standing position. Subjects perform this task 5 times and data is presented as their faster time.
Time Frame: baseline
Measure: Number; unit: seconds
Arm/Group | Placebo | Testosterone
Number analyzed (Participants) | 1 | 1
seconds | 1.08 | 2.02

13. Secondary Outcome: Chair Raise as Measured by Short Physical Performance Battery (SPPB) at 10 Weeks
Description: During the chair rise section of the Short Physical Performance Battery (SPPB), subjects are timed while they rise from a seated (chair) to standing position. Subjects perform this task 5 times and data is presented as their best time.
Time Frame: 10 Weeks
Measure: Number; unit: seconds
Arm/Group | Placebo | Testosterone
Number analyzed (Participants) | 1 | 1
seconds | 1.08 | 1.01

ADVERSE EVENTS:
Time Frame: 10 weeks
Arm/Group | Placebo | Testosterone
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No